CLINICAL TRIAL: NCT00936260
Title: Drug Holidays in the Treatment With Alendronate in Postmenopausal Women With Osteoporosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ciudad Universitaria, Spain (Other)
Responsible Party: Esther Alvarez-Rodriguez, University San Carlos Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: individual reseacher
Record Dates: First submitted 2009-07-09; First posted 2009-07-10 (Estimated); Last update posted 2009-07-10 (Estimated); Status verified 1998-01

CONDITIONS: Osteoporosis
Keywords: osteoporosis; postmenopausal; alendronate
MeSH Terms: conditions — Osteoporosis | interventions — Alendronate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (8):
- alendronate 6 years (Experimental)
  Interventions: Drug: alendronate
- alendronate 5 years (Experimental): No treatment during year 6th
  Interventions: Drug: alendronate
- alendronate 5 years, not continued (Experimental): No treatment during year 5th
  Interventions: Drug: alendronate
- alendronate 4 years (Experimental): No treatment during year 5th and 6th
  Interventions: Drug: alendronate
- alendronate 5 years, uncontinued (Experimental): No treatment during year 4th
  Interventions: Drug: alendronate
- alendronate 4 years, not continued (Experimental): No treatment during year 4th and 6th
  Interventions: Drug: alendronate
- alendronate 4 years, uncontinued (Experimental): No treatment during year 4th and 5th
  Interventions: Drug: alendronate
- Alendronato 3 years (Experimental): No treatment during the last 3 years
  Interventions: Drug: alendronate

INTERVENTIONS:
Drug: alendronate — several duration of treatment
  Other Names: fosamax

SUMMARY:
The purpose of this study is to determine the duration of the treatment with alendronate in postmenopausal women with osteoporosis.

DETAILED DESCRIPTION:
The duration of the treatment with alendronate is not well established. The investigators recruited 228 women with postmenopausal osteoporosis. They all received alendronate during the first 3 years of monitoring and were later on randomized to whether different regimens of intermittent treatment or to carry on 3 years more.

ELIGIBILITY:
Inclusion Criteria:

* postmenopausal osteoporosis under densitometric criteria of the World Health Organization

Exclusion Criteria:

* secondary osteoporosis
* alteration in analytic parameters (total proteins, calcium, phosphorus, vitamin D, parathyroid hormone, thyroid hormone, transaminase, creatinine)

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 228 (Actual)
Dates: Start 1998-01; Primary Completion 2004-12 (Actual); Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
Bone mineral density | Every year

SECONDARY OUTCOMES:
Fractures | Every year

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Lozano Tonkin, doctor, Study Director — university san carlos hospital
Locations (1):
- University San Carlos Hospital, Madrid, Madrid, Spain